CLINICAL TRIAL: NCT02446899
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Phase 3 Study Evaluating the Efficacy and Safety of Anifrolumab in Adult Subjects With Active Systemic Lupus Erythematosus
Brief Title: Efficacy and Safety of Anifrolumab Compared to Placebo in Adult Subjects With Active Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3461C00004
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Active Systemic Lupus Erythematosus
Keywords: Active Systemic Lupus Erythematosus
MeSH Terms: interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anifrolumab (Experimental): Anifrolumab 300 mg intravenous infusion (IV) administered every 4 weeks for a total of 13 doses.
  Interventions: Biological: Anifrolumab
- Placebo (Placebo Comparator): Placebo intravenous infusion (IV) administered every 4 weeks for a total of 13 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Anifrolumab — Intravenous infusion (IV)
  Arms: Anifrolumab
Drug: Placebo — Intravenous infusion (IV)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of an intravenous treatment regimen of anifrolumab versus placebo in adult participants with moderately to severely active, autoantibody-positive systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This is a Phase 3, multicentre, multinational, randomised, double-blind, placebo-controlled study to evaluate the efficacy and safety of an intravenous treatment regimen of anifrolumab versus placebo in participants with moderately to severely active, autoantibody-positive systemic lupus erythematosus (SLE) while receiving standard of care (SOC) treatment. Participants must be taking either 1 or any combination of the following: oral corticosteroids (OCS), antimalarial, and/or immunosuppressants. The study will be performed in adult participants aged 18 to 70 years of age.

Approximately 360 participants receiving SOC treatment will be randomised in a 1:1 ratio to receive a fixed intravenous dose of anifrolumab 300 mg or placebo every 4 weeks for a total of 13 doses (Week 0 to Week 48), with the primary endpoint evaluated at the Week 52 visit. Investigational product will be administered as an intravenous infusion (IV) via an infusion pump over a minimum of 30 minutes, every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 through 70 years at the time of screening
2. Diagnosis of paediatric or adult SLE with a diagnosis of SLE according to the ACR 1982 revised criteria ≥24 weeks prior to signing the Informed Consent form (ICF)
3. Currently receiving at least 1 of the following:

   1. Where prednisone is the single standard of care medication (ie, the subject is not concurrently receiving any medication listed in inclusion criterion 3(c)), a dose of oral prednisone ≥7.5 mg/day but ≤40 mg/day (or prednisone equivalent) for a minimum of 8 weeks prior to Day 1. In addition, the dose of oral prednisone or prednisone equivalent the subject is taking must be stable for a minimum of 2 weeks prior to randomisation
   2. Where prednisone is not the single standard of care medication (ie, the subject is concurrently receiving at least one medication listed in inclusion criterion 3(c), a dose of oral prednisone (≤40 mg/day) (or prednisone equivalent) for a minimum of 2 weeks prior to signing of the ICF. In addition, the dose of oral prednisone or prednisone equivalent the subject is taking must be stable for a minimum of 2 weeks prior to randomisation.
   3. Any of the following medications administered for a minimum of 12 weeks prior to signing the informed consent, and at a stable dose for a minimum of 8 weeks prior to signing the informed consent and through Day 1:

   (i) Azathioprine ≤200 mg/day (ii) Antimalarial (eg, chloroquine, hydroxychloroquine, quinacrine) (iii) Mycophenolate mofetil ≤2 g/day or mycophenolic acid ≤1.44 g/day (iv) Oral, subcutaneous (SC), or intramuscular methotrexate ≤25 mg/week (v) Mizoribine ≤150 mg/day
4. Fulfils at least 4 of the 11 ACR modified 1982 classification criteria for SLE, at least 1 of which must be:

   1. Positive antinuclear antibody (ANA) test at screening by immunofluorescent assay (IFA) at the central laboratory with titre ≥1:80; OR
   2. Anti-dsDNA antibodies at screening elevated to above normal (including indeterminate), as per the central laboratory; OR
   3. Anti-Smith (anti-Sm) antibody at screening elevated to above normal as per the central laboratory
5. At Screening, Disease Activity Adjudication Group confirmation of:

   SLEDAI-2K Criteria: SLEDAI-2K score ≥6 points and "Clinical" SLEDAI-2K score ≥4 points. The "Clinical" SLEDAI-2K is the SLEDAI-2K assessment score without the inclusion of points attributable to any urine or laboratory results including immunologic measures.
6. Must not have active or latent TB on either chest radiograph or by quantiferon gold test
7. Day 1 "Clinical" SLEDAI-2K score ≥4 points
8. OCS dose stable for at least 2 weeks prior to randomisation
9. Stable SLE SOC treatment at the time of randomisation
10. Women of child-bearing potential must have a negative serum β-hCG test at and negative urine pregnancy test at randomisation prior to administration of investigational product

Exclusion Criteria:

1. Receipt of any investigational product (small molecule or biologic agent) within 4 weeks or 5 half-lives prior to signing of the ICF, whichever is greater
2. Receipt of any of the following:

   (a) Intra-articular, intramuscular or IV glucocorticosteroids within 6 weeks prior to Day 1
3. History of, or current diagnosis of, a clinically significant non SLE-related vasculitis syndrome.
4. Active severe or unstable neuropsychiatric SLE
5. Active severe SLE-driven renal disease
6. Diagnosis (within 1 year of signing the ICF) of mixed connective tissue disease or any history of overlap syndromes of SLE or SSc.
7. History of, or current, inflammatory joint or skin disease other than SLE
8. History of any non-SLE disease that has required treatment with oral or parenteral corticosteroids for more than 2 weeks within the last 24 weeks prior to signing the ICF
9. 26.27. Known history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the subject to infection, or a positive result for human immunodeficiency virus (HIV) infection confirmed by central laboratory at screening. Subjects refusing HIV testing during the screening period will not be eligible for study participation
10. Confirmed positive test for hepatitis B or hepatitis C
11. Any severe herpes infection at any time prior to Week 0 (Day 1)
12. Opportunistic infection requiring hospitalisation or intravenous antimicrobial treatment within 3 years prior to randomization
13. History of cancer, apart from:

    1. Squamous or basal cell carcinoma of the skin that has been successfully treated
    2. Cervical cancer in situ that has been successfully treated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lilia Pineda, MD, Study Director — Medical Science Director
Locations (99):
- United States (31):
  - Research Site, Covina, California
  - Research Site, Hemet, California
  - Research Site, Los Angeles, California
  - Research Site, San Leandro, California
  - Research Site, Torrance, California
  - Research Site, Upland, California
  - Research Site, Denver, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Brandon, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Cruces, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Stafford, Texas
  - Research Site, Arlington, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
- Argentina (3):
  - Research Site, Buenos Aires
  - Research Site, Mendoza
  - Research Site, Quilmes
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Merksem
- Brazil (3):
  - Research Site, Goiânia
  - Research Site, Juiz de Fora
  - Research Site, São Paulo
- Research Site, Plovdiv, Bulgaria
- Canada (2):
  - Research Site, Hamilton, Ontario
  - Research Site, Rimouski, Quebec
- France (6):
  - Research Site, Bordeaux
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Toulouse
- Germany (5):
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Jena
  - Research Site, Mainz
  - Research Site, München
- Japan (15):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kitakyushu-shi
  - Research Site, Kurashiki-shi
  - Research Site, Meguro-ku
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Omura-shi
  - Research Site, Sapporo
  - Research Site, Sasebo-shi
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Tsukuba
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Klaipėda
- Mexico (7):
  - Research Site, Chihuahua City
  - Research Site, León
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Morelia
  - Research Site, San Luis Potosí City
- Russia (6):
  - Research Site, Kemerovo
  - Research Site, Petrozavodsk
  - Research Site, Smolensk
  - Research Site, Tolyatti
  - Research Site, Vladimir
  - Research Site, Yaroslavl
- South Africa (3):
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Stellenbosch
- South Korea (3):
  - Research Site, Jeju City
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (8):
  - Research Site, Barcelona
  - Research Site, Getafe
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Mérida
  - Research Site, Santiago de Compostela
  - Research Site, Servilla
  - Research Site, Vigo

REFERENCES:
- [Derived] Morand EF, Abreu G, Furie RA, Golder V, Tummala R. Lupus low disease activity state attainment in the phase 3 TULIP trials of anifrolumab in active systemic lupus erythematosus. Ann Rheum Dis. 2023 May;82(5):639-645. doi: 10.1136/ard-2022-222748. Epub 2023 Jan 23. PMID 36690388
- [Derived] Bruce IN, van Vollenhoven RF, Morand EF, Furie RA, Manzi S, White WB, Abreu G, Tummala R. Sustained glucocorticoid tapering in the phase 3 trials of anifrolumab: a post hoc analysis of the TULIP-1 and TULIP-2 trials. Rheumatology (Oxford). 2023 Apr 3;62(4):1526-1534. doi: 10.1093/rheumatology/keac491. PMID 36018235
- [Derived] Bruce IN, Furie RA, Morand EF, Manzi S, Tanaka Y, Kalunian KC, Merrill JT, Puzio P, Maho E, Kleoudis C, Albulescu M, Hultquist M, Tummala R. Concordance and discordance in SLE clinical trial outcome measures: analysis of three anifrolumab phase 2/3 trials. Ann Rheum Dis. 2022 Jul;81(7):962-969. doi: 10.1136/annrheumdis-2021-221847. Epub 2022 May 17. PMID 35580976
- [Derived] Vital EM, Merrill JT, Morand EF, Furie RA, Bruce IN, Tanaka Y, Manzi S, Kalunian KC, Kalyani RN, Streicher K, Abreu G, Tummala R. Anifrolumab efficacy and safety by type I interferon gene signature and clinical subgroups in patients with SLE: post hoc analysis of pooled data from two phase III trials. Ann Rheum Dis. 2022 Jul;81(7):951-961. doi: 10.1136/annrheumdis-2021-221425. Epub 2022 Mar 25. PMID 35338035
- [Derived] Loncharich MF, Anderson CW. Interferon Inhibition for Lupus with Anifrolumab: Critical Appraisal of the Evidence Leading to FDA Approval. ACR Open Rheumatol. 2022 Jun;4(6):486-491. doi: 10.1002/acr2.11414. Epub 2022 Feb 14. PMID 35157371
- [Derived] Chia YL, Zhang J, Tummala R, Rouse T, Furie RA, Morand EF. Relationship of anifrolumab pharmacokinetics with efficacy and safety in patients with systemic lupus erythematosus. Rheumatology (Oxford). 2022 May 5;61(5):1900-1910. doi: 10.1093/rheumatology/keab704. PMID 34528084
- [Derived] Furie R, Morand EF, Askanase AD, Vital EM, Merrill JT, Kalyani RN, Abreu G, Pineda L, Tummala R. Anifrolumab reduces flare rates in patients with moderate to severe systemic lupus erythematosus. Lupus. 2021 Jul;30(8):1254-1263. doi: 10.1177/09612033211014267. Epub 2021 May 12. PMID 33977796
- [Derived] Furie R, Morand EF, Bruce IN, Isenberg D, van Vollenhoven R, Abreu G, Pineda L, Tummala R. What Does It Mean to Be a British Isles Lupus Assessment Group-Based Composite Lupus Assessment Responder? Post Hoc Analysis of Two Phase III Trials. Arthritis Rheumatol. 2021 Nov;73(11):2059-2068. doi: 10.1002/art.41778. Epub 2021 Sep 22. PMID 33913260
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Morand EF, Furie R, Tanaka Y, Bruce IN, Askanase AD, Richez C, Bae SC, Brohawn PZ, Pineda L, Berglind A, Tummala R; TULIP-2 Trial Investigators. Trial of Anifrolumab in Active Systemic Lupus Erythematosus. N Engl J Med. 2020 Jan 16;382(3):211-221. doi: 10.1056/NEJMoa1912196. Epub 2019 Dec 18. PMID 31851795
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461C00004&attachmentIdentifier=3a779c1e-b522-4240-8d7f-fd4e6848a9d1&fileName=D3461C00004_CSP_redactions_applied.pdf&
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461C00004&attachmentIdentifier=c6a17786-1293-46c9-87e6-d6dda2c86d2a&fileName=D3461C00004_Redacted_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the trial at 119 sites in 15 countries worldwide.
Pre-assignment Details: 8 participants were assigned study drug, but due to non-compliance were analyzed separately (not included in the participant flow). 3 additional participants were assigned study drug & included in the participant flow, but did not receive study drug due to an adverse event (1 Anifrolumab 300mg) & failure to meet randomization criteria (2 Placebo).
Groups:
- Anifrolumab 300 mg: Anifrolumab (300 mg) administered via an intravenous infusion (IV) every 4 weeks for up to 48 weeks (13 doses).
- Placebo: Matching placebo administered via an intravenous infusion (IV) every 4 weeks for up to 48 weeks (13 doses).
Period: Overall Study
Arm/Group | Anifrolumab 300 mg | Placebo
Started | 181 | 184
Received Study Drug | 180 | 182
Completed | 156 | 136
Not Completed | 25 | 48
Not completed — Adverse Event | 4 | 7
Not completed — Condition Under Investigation Worsened | 1 | 4
Not completed — Study Specific Withdrawal Criteria | 1 | 0
Not completed — Lack of Efficacy | 2 | 8
Not completed — Lost to Follow-up | 1 | 3
Not completed — Severe Non-Compliance to Protocol | 0 | 1
Not completed — Withdrawal by Subject | 11 | 19
Not completed — Miscellaneous | 5 | 4
Not completed — Failure to Meet Randomization Criteria | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set: All participants who were randomized and received at least one dose of the study drug. 3 participants discontinued the study prior to receiving the study drug and are not included in the full analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anifrolumab 300 mg | Placebo | Total
Number analyzed (Participants) | 180 | 182 | 362
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 175 | 181 | 356
  >=65 years | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (11.95) | 41.1 (11.47) | 42.1 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 170 | 338
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 54 | 108
  Not Hispanic or Latino | 118 | 120 | 238
  Unknown or Not Reported | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 110 | 107 | 217
  Black or African American | 17 | 25 | 42
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 4 | 1 | 5
  Other | 11 | 11 | 22
  Missing | 8 | 8 | 16
Geographic region [Count of Participants; unit: Participants]
  Asia Pacific | 27 | 26 | 53
  Europe | 51 | 46 | 97
  Latin America | 35 | 32 | 67
  United States/Canada | 64 | 68 | 132
  Rest of World (South Africa) | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved the British Isles Lupus Assessment Group Based Composite Lupus Assessment (BICLA) Response at Week 52
Description: Composite endpoint BICLA was defined by meeting all of the following criteria:
  * Reduction of all baseline British Isles Lupus Assessment Group (BILAG)-2004 A to B/C/D and baseline BILAG-2004 B to C/D, and no BILAG-2004 worsening in other organ systems, as defined by ≥1 new BILAG-2004 A or ≥2 new BILAG-2004 B
  * No worsening from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K), where worsening is defined as an increase from baseline of >0 points in SLEDAI-2K
  * No worsening from baseline in participants' lupus disease activity, where worsening is defined by an increase ≥0.30 points on a 3-point Physician's Global Assessment (PGA) visual analogue scale (VAS)
  * No discontinuation of investigational product
  * No use of restricted medications beyond the protocol allowed threshold before assessment
Time Frame: Baseline; Week 52
Population: Full Analysis Set: All participants who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 180 | 182
Participants | 86 | 57
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Test type: Superiority — The difference in estimates and associated 95% CI are weighted and are calculated using a stratified Cochran-Mantel-Haenszel (CMH) approach, with stratification factors (SLEDAI-2K score at screening [<10 points vs >= 10 points], Week 0 OCS dose [<10 mg/day vs >=10 mg/day prednisone or equivalent] and type I IFN gene signature test result at screening [high vs low]); p = 0.0013, Cochran-Mantel-Haenszel — Nominal p-value; Mean Difference (Final Values) = 16.3, 95% CI 2-sided [6.3 to 26.3]

2. Secondary Outcome: Number of Participants Who Achieved the British Isles Lupus Assessment Group Based Composite Lupus Assessment (BICLA) Response at Week 52 in the IFN Test-High Sub-group
Description: Defined by meeting all of the following criteria:
  * Reduction of all baseline British Isles Lupus Assessment Group (BILAG)-2004 A to B/C/D and baseline BILAG-2004 B to C/D, and no BILAG-2004 worsening in other organ systems, as defined by ≥1 new BILAG-2004 A or ≥2 new BILAG-2004 B
  * No worsening from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K), where worsening is defined as an increase from baseline to >0 points in SLEDAI-2K
  * No worsening from baseline in participants' lupus disease activity, where worsening is defined by an increase ≥0.30 points on a 3-point Physician's Global Assessment (PGA) visual analogue scale (VAS)
  * No discontinuation of investigational product
  * No use of restricted medications beyond the protocol allowed threshold before assessment
Time Frame: Baseline; Week 52
Population: Full Analysis Set: All participants who were randomized and received at least one dose of study drug, with a high interferon (IFN) test result at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 150 | 151
Participants | 72 | 46
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; The difference in estimates and associated 95% CI are weighted and are calculated using a stratified Cochran-Mantel-Haenszel (CMH) approach, with stratification factors (SLEDAI-2K score at screening [<10 points vs >= 10 points], Week 0 OCS dose [<10 mg/day vs >=10 mg/day prednisone or equivalent] and type I IFN gene signature test result at screening [high vs low]); Test type: Superiority; p = 0.0022, Cochran-Mantel-Haenszel — Adjusted p-value; Mean Difference (Final Values) = 17.3, 95% CI 2-sided [6.5 to 28.2]

3. Secondary Outcome: Number of Participants Who Achieved and Maintained an Oral Corticosteroids (OCS) Dose of ≤7.5 mg/Day at Week 52 in the Sub-Group of Participants With Baseline OCS ≥10 mg/Day
Description: Maintained OCS reduction was defined by meeting all of the following criteria:
  * Achieve an OCS dose of ≤7.5 mg/day prednisone or equivalent by Week 40
  * Maintain an OCS dose ≤7.5 mg/day prednisone or equivalent from Week 40 to Week 52
  * No discontinuation of investigational product
  * No use of restricted medications beyond the protocol allowed threshold before assessment
Time Frame: Week 40; Week 52
Population: Full Analysis Set: All participants who were randomized and received at least one dose of study drug, who had a baseline OCS dose of ≥10 mg/day.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 87 | 83
Participants | 45 | 25
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0135, Cochran-Mantel-Haenszel — Adjusted p-value; Mean Difference (Final Values) = 21.2, 95% CI 2-sided [6.8 to 35.7]

4. Secondary Outcome: Number of Participants With a ≥50% Reduction in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score at Week 12 in The Sub-Group of Participants With Baseline CLASI Activity Score of ≥10
Description: 50% reduction in CLASI activity score compared to baseline was defined by meeting all of the following criteria:
  * Achieve ≥50% reduction of CLASI activity score at Week 12 compared to baseline
  * No discontinuation of investigational product
  * No use of restricted medications beyond the protocol allowed threshold before assessment
Time Frame: Baseline; Week 12
Population: Full Analysis Set: All participants who were randomized and received at least one dose of study drug, and who had a CLASI activity score of ≥10 at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 49 | 40
Participants | 24 | 10
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0392, Cochran-Mantel-Haenszel — Adjusted p-value; Mean Difference (Final Values) = 24.0, 95% CI 2-sided [4.3 to 43.6]

5. Secondary Outcome: Number of Participants With ≥50% Reduction in Joint Counts at Week 52 in The Sub-group of Participants With ≥6 Swollen and ≥6 Tender Joints at Baseline
Description: 50% reduction in the number of swollen and tender joints compared to baseline was defined by meeting all of the following criteria:
  * Achieve ≥50% reduction from baseline in the number of swollen and tender joints, separately
  * No discontinuation of investigational product
  * No use of restricted medications beyond the protocol allowed threshold before assessment
Time Frame: Baseline; Week 52
Population: Full Analysis Set: All participants who were randomized and received at least one dose of study drug, and who had ≥6 swollen and ≥6 tender joints at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 71 | 90
Participants | 30 | 34
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5469, Cochran-Mantel-Haenszel — Adjusted p-value; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-10.6 to 20.0]

6. Secondary Outcome: Annualised Flare Rate Through 52 Weeks
Description: A flare was defined as either 1 or more new British Isle Lupus Assessment Group (BILAG-2004) A or 2 or more new BILAG-2004 B items compared to the previous visit. The occurrence of a new flare was checked for each available visit versus the previous available visit up to Week 52. If no new flares occurred, the number of flares was set to 0. Otherwise all flares were counted leading to the maximum number of flares of 13. The annualized flare rate was calculated as the number of flares divided by the flare exposure time in days multiplied with 365.25 (1 year). The flare exposure time is the time up to Week 52 (date of BILAG-2004 assessment at Week 52) or up to the date of last available BILAG-2004 assessment.
Time Frame: Baseline to Week 52
Population: Full Analysis Set: All participants who were randomized and received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Annualized flare rate ratio
Arm/Group | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 180 | 182
Annualized flare rate ratio | 0.43 [0.31 to 0.59] | 0.64 [0.47 to 0.86]
Statistical Analysis 1: Comparison: Anifrolumab 300 mg vs Placebo; Analysed using a negative binomial regression model. The response variable in the model is the number of flares over the 52-week treatment period. The model includes covariates of treatment group, and the stratification factors (SLEDAI-2K score at screening [<10 points vs >=10 points], Week 0 OCS dose [<10 mg/day vs >=10 mg/day prednisone or equivalent] and type I IFN gene signature test result at screening [high vs low]). The logarithm of the follow-up time is used as an offset variable; Test type: Superiority; p = 0.0809, Negative binomial regression — Adjusted p-value; Rate Ratio = 0.67, 95% CI 2-sided [0.48 to 0.94]

7. Secondary Outcome: Number of Participants With One or More Adverse Events (AEs)
Description: An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. AEs were collected throughout the duration of the study, from baseline until end of follow-up (a maximum of 12 weeks post last dose [Week 48]), or until Week 52 for participants who enrolled onto the long term extension (LTE). The reported value is inclusive of serious and non-serious AEs.
Time Frame: Baseline to end of study (Maximum of 60 weeks)
Population: Full Analysis Set: All participants who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 180 | 182
Participants | 162 | 154

8. Secondary Outcome: Number of Participants With One or More Adverse Events of Special Interest (AESIs)
Description: An AESI is an adverse event (AE) of scientific and medical concern specific to understanding biologics. An AESI may be serious or non-serious. AESI are serious infections, including non-opportunistic serious infections, opportunistic infections, anaphylaxis, malignancy, herpes zoster, tuberculosis (TB) (including latent TB), influenza, vasculitis (non-systemic lupus erythematosus [SLE]), and major adverse cardiovascular events (MACE) (including stroke, myocardial infarction [MI], or cardiovascular death).
  AESIs were collected throughout the study, from baseline until end of follow-up (a maximum of 12 weeks post last dose [Week 48]), or until Week 52 for participants who enrolled onto the long term extension (LTE).
Time Frame: Baseline to end of study (Maximum of 60 weeks)
Population: Full Analysis Set: All participants who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 180 | 182
Participants | 29 | 20

9. Secondary Outcome: Number of Participants With a Potentially Clinically Important Change From Baseline in Vital Sign Measurements
Description: Vital sign measurements included oral temperature, blood pressure (BP), pulse rate, and respiratory rate.
  Vital signs were collected throughout the duration of the study, from baseline until end of follow-up (a maximum of 12 weeks post last dose [Week 48]), or until Week 52 for participants who enrolled onto the long term extension (LTE).
Time Frame: Baseline to end of study (Maximum of 60 weeks)
Population: Full Analysis Set: All participants who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 180 | 182
Participants | 45 | 45

10. Secondary Outcome: Number of Participants With a Potentially Clinically Important Change From Baseline in Clinical Laboratory Tests
Description: Clinical laboratory tests were analyzed in a central clinical laboratory and included hematology, serum chemistry and urinalysis tests.
  Laboratory values were collected throughout the duration of the study, from baseline until end of follow-up (a maximum of 12 weeks post last dose [Week 48]), or until Week 52 for participants who enrolled onto the long term extension (LTE).
Time Frame: Baseline to end of study (Maximum of 60 weeks)
Population: Full Analysis Set: All participants who were randomized and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Anifrolumab 300 mg | Placebo
Number analyzed (Participants) | 180 | 182
Participants | 72 | 87

ADVERSE EVENTS:
Time Frame: Day 1 to end of study (Maximum of 60 weeks)
Description: AEs were either spontaneously reported by the participant or reported in response to open questions, revealed by observation, or were changes from baseline/deterioration in tests and vital signs that met serious adverse event (SAE) criteria or led to study drug discontinuation. A treatment-emergent adverse event (TEAE) is defined as an AE with an onset that occurs after receiving study drug.
  Full analysis set: All participants who had received at least one dose of study drug.
Arm/Group | Anifrolumab 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/180 | 0/182
Serious Adverse Events (participants affected / at risk) | 16/180 | 34/182
Other Adverse Events (participants affected / at risk) | 125/180 | 99/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anifrolumab 300 mg (N=180) | Placebo (N=182)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Chilaiditi's syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 7 (7)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anifrolumab 300 mg (N=180) | Placebo (N=182)
Nausea (Gastrointestinal disorders) | 7 (7) | 10 (11)
Bronchitis (Infections and infestations) | 23 (31) | 8 (8)
Herpes zoster (Infections and infestations) | 12 (12) | 3 (3)
Nasopharyngitis (Infections and infestations) | 28 (42) | 23 (31)
Sinusitis (Infections and infestations) | 13 (21) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 42 (57) | 19 (24)
Urinary tract infection (Infections and infestations) | 21 (27) | 26 (40)
Infusion related reaction (Injury, poisoning and procedural complications) | 25 (42) | 14 (27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 3 (3)
Headache (Nervous system disorders) | 11 (13) | 18 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT02446899/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT02446899/SAP_001.pdf